CLINICAL TRIAL: NCT05397574
Title: Intraoperative Hyperspectral Imaging for Real-time Fluorescence-guided Surgery of Low Grade Glioma
Brief Title: Intraoperative Hyperspectral Imaging for Fluorescence Guided Surgery in Low Grade Gliomas
Acronym: Neuro-qFHSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 307291
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Neurosurgery; Neuro-Oncology; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to obtain images of brain tumours during surgery using a new type of surgical camera. The study will assess how the information obtained from the images during surgery matches the removed tissue. Data will also be used to develop the system's key computer-processing features. This will enable real-time information to be given to the surgeon whilst they are performing the procedure and has the potential to make neurosurgery safer and more precise.

DETAILED DESCRIPTION:
High grade gliomas (HGG) and low grade gliomas (LGG) are the commonest CNS cancers, with LGGs accounting for 6.4% of all adult cases (Ostrom 2019). Despite LGGs typically being slow-growing, over 70% of them transform into higher-grade tumours or become aggressive within a decade (Jooma 2019). Median survival for LGG patients spans 5.6 to 13.3 years (Brown 2019). Gross total resection (GTR) improves 5-year LGG survival rates from 60% to 90% when compared to subtotal resection. However, GTR (>96% tumour removal) is frequently not achieved because despite advanced techniques being available, surgeons are unable to clearly visualise the tumour and its boundaries in real-time during surgery.

There is an acute need to improve outcomes for affected brain tumour patients. Patients undergoing surgery have significantly improved outcomes and increased life expectancy if complete tumour removal is achieved. However, close to 30% of patients are left with residual tumour tissue after surgery. Successful surgery indeed mandates maximal safe tumour removal: surgeons need to avoid damaging sensitive areas that undertake vital functions and preserve crucial nerves and blood vessels. Even with the most advanced current techniques, it is not possible to always identify tumour and critical structures reliably during surgery. Furthermore, because one cannot objectively measure the blood supply and oxygenation of brain tissue during surgery, it is difficult to judge if injury is being caused during the operation.

To address the pressing clinical need of improved surgical precision and patient safety during low grade glioma surgery, we aim to develop an imaging system capable of quantitative wide-field fluorescence imaging for seamless real-time surgical guidance. This project aims to improve patient survival by delivering a precise assistive tool for neurosurgeons performing LGG surgery by evaluating this device in patients undergoing glioma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and over
* Patients with a diagnosis of a probable glioma (any grade), who are scheduled for elective surgery
* Patients able to provide written informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients who have previously had brain surgery
* Patients unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioma surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of qFHSI data with histological analysis of the corresponding biopsied pathological tissue | 6-12 months
  To correlate ex vivo and in vivo qFHSI data with histological analysis of the corresponding biopsied glioma tissue

SECONDARY OUTCOMES:
Safety of qFHSI in surgery | 24-36 months
  To demonstrate safety of our intraoperative qFHSI device during glioma surgery
Tissue diagnosis | 24 months
  To collect ex vivo and in vivo qFHSI data during glioma surgery for tissue analysis, algorithmic development and testing
Accuracy of biophotonics algorithm | 24-36 months
  To evaluate accuracy of the computational biophotonics algorithm to determine 5-ALA-PpIX concentration in imaged tissue
Qualitative assessment | 24-36 months
  A qualitative assessment of the impact that using the device has on surgical workflow

CONTACTS AND LOCATIONS:
Locations (1):
- King's College NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided